CLINICAL TRIAL: NCT07150299
Title: Myocardial Perfusion Changes Following Optimal Medical Treatment in Symptomatic Hypertrophic Cardiomyopathy
Acronym: oHCM
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel Dalos, Chief resident, Medical University of Vienna
Other Study IDs: CV027-1201; 1492/2025 (Other: Medical University of Vienna)
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM)
Keywords: Myocardial Perfusion
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mavacamten in clinical routine use — Clinical observation of mavacamten use

SUMMARY:
Background: Microvascular dysfunction is a hallmark of hypertrophic obstructive cardiomyopathy (HOCM) and can be visualized non-invasively using cardiac magnetic resonance (CMR) perfusion imaging. In parallel, the six-minute walk test (6MWT) is an established clinical tool to assess submaximal exercise capacity in patients with structural heart disease. Despite its widespread use, the relationship between objective changes in myocardial perfusion and functional improvements assessed by the 6MWT remains insufficiently explored in patients with HOCM on optimal medical therapy (OMT).

Aim:This study aims to evaluate whether changes in functional capacity, measured by the 6MWT, correlate with changes in myocardial perfusion reserve (MPR) in HOCM patients treated with OMT.

Methods: We will include patients diagnosed with obstructive HCM who previously underwent clinically indicated CMR perfusion scans for risk stratification. These patients are regularly followed in the HCM outpatient clinic of the Medical University of Vienna, where standardized 6MWTs are performed in routine care. Approximately one year after the baseline CMR, a follow-up CMR will be conducted to assess changes in perfusion parameters. This second CMR is clinically justified for improved individual risk stratification as recommended by the 2023 ESC Guidelines on Cardiomyopathies.

The primary objective is to assess the correlation between the change in the walking distance in the 6MWT and the change in MPR over a one-year interval. Secondary endpoints include changes in myocardial blood flow (MBF) at rest and during pharmacological stress. All assessments will be integrated with clinical, echocardiographic, and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Willingness to provide written informed consent
* Diagnosis of obstructive HCM based on ESC 2023 criteria
* Planned CMR with myccardial perfusion for clinical purposes
* Receiving guideline-conform OMT
* Ability and willingness to undergo follow-up imaging and testing
* Written informed consent

Exclusion Criteria:

* Claustrophobia or other contraindication for CMR imaging
* Significant coronary artery disease and/or prior stent implantation or coronary artery bypass graft surgery
* History of sudden cardiac arrest or sustained ventricular arrhythmia 12 months prior to screening
* Glomerular filtration rate < 30ml/min/m2
* Significant hepatic impairment defined as 3x upper limit of normal of transaminases, total bilirubin, or alkaline phosphatase; hepatic cirrhosis
* Known allergy to contrast agent
* Alternative disease causing hypertrophic cardiomyopathy (e.g. cardiac amyloidosis, Morbus Fabry)
* Pregnant women (and women with childbearing potential with desire for pregnancy)
* Breastfeeding women
* Unwillingness to comply with the study protocol and its procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oHCM on maximal tolerated background therapy which will receive mavacamten as add-on
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between myocardial perfusion reserve changes and changes in the performed distance in 6MWT. | One year of maximal tolerated dose of mavacamten
  Correlation between myocardial perfusion reserve changes and changes in the performed distance in 6MWT.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT07150299/Prot_000.pdf